CLINICAL TRIAL: NCT05523089
Title: A Proof-of-concept, Randomized, Double-blind, Placebo-controlled, Phase 2a Study to Assess the Prophylactic Antiviral Activity Against Influenza, Safety, Tolerability, and Pharmacokinetics of CD388 Via a Human Viral Challenge Model
Brief Title: The Effectiveness of CD388 to Prevent Flu in an Influenza Challenge Model in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CD388.SQ.2.02
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Placebo (Arm 1) (Placebo Comparator): In Cohort 1, up to 30 participants will be randomized to receive a single dose of placebo, administered by subcutaneous (SQ) injection, prior to being inoculated with the influenza challenge virus. Based on an interim analysis to be performed on data collected from the evaluation of Cohort 1 participants who have completed the inpatient phase at the time the interim analysis is performed, additional participants (of a number to be informed by the interim analysis) may be randomized into Cohort 2 in an extension of this Arm 1, to receive a single dose of placebo by SQ injection prior to viral challenge.
  Interventions: Drug: Saline placebo
- CD388 High Dose (Arm 2) (Experimental): In Cohort 1, up to 30 participants will be randomized to receive a single dose of 150 milligrams (mg) CD388, administered by SQ injection, prior to being inoculated with the influenza challenge virus. Based on an interim analysis to be performed on data collected from the evaluation of Cohort 1 participants who have completed the inpatient phase at the time the interim analysis is performed, additional participants (of a number to be informed by the interim analysis) may be randomized into Cohort 2 in an extension of this Arm 2, to receive a single dose of 150 mg CD388 by SQ injection prior to viral challenge.
  Interventions: Combination Product: CD388
- CD388 Low Dose 1 (Arm 3) (Experimental): In Cohort 1, up to 30 participants will be randomized to receive a single dose of 50 mg CD388, administered by SQ injection, prior to being inoculated with the influenza challenge virus. Based on an interim analysis to be performed on data collected from the evaluation of Cohort 1 participants who have completed the inpatient phase at the time the interim analysis is performed, additional participants (of a number to be informed by the interim analysis) may be randomized into Cohort 2 in an extension of this Arm 3, to receive a single dose of 50mg CD388 by SQ injection prior to viral challenge.
  Interventions: Combination Product: CD388
- CD388 Low Dose 2 (Optional Arm 4) (Experimental): Based on an interim analysis to be performed on data collected from the evaluation of Cohort 1 participants who have completed the inpatient phase at the time the interim analysis is performed, participants (of a number to be informed by the interim analysis) may be randomized into Cohort 2 in this Optional Arm 4, to receive a single dose of CD388 lower than 150 mg (TBD based on PK results obtained in the first-in-human study CD388.IM.SQ.1.01, as well as the interim analysis), administered by SQ injection, prior to being inoculated with the influenza challenge virus.
  Interventions: Combination Product: CD388
- CD388 Low Dose 3 (Optional Arm 5) (Experimental): Based on an interim analysis to be performed on data collected from the evaluation of Cohort 1 participants who have completed the inpatient phase at the time the interim analysis is performed, participants (of a number to be informed by the interim analysis) may be randomized into Cohort 2 in this Optional Arm 5, to receive a single dose of CD388 lower than 150 mg (TBD based on PK results obtained in the first-in-human study CD388.IM.SQ.1.01, as well as the interim analysis), administered by SQ injection, prior to being inoculated with the influenza challenge virus.
  Interventions: Combination Product: CD388
- CD388 Low Dose 4 (Optional Arm 6) (Experimental): Based on an interim analysis to be performed on data collected from the evaluation of Cohort 1 participants who have completed the inpatient phase at the time the interim analysis is performed, participants (of a number to be informed by the interim analysis) may be randomized into Cohort 2 in this Optional Arm 6, to receive a single dose of CD388 lower than 150 mg (TBD based on PK results obtained in the first-in-human study CD388.IM.SQ.1.01, as well as the interim analysis), administered by SQ injection, prior to being inoculated with the influenza challenge virus.
  Interventions: Combination Product: CD388

INTERVENTIONS:
Drug: Saline placebo — Sterile normal saline for injection
  Arms: Placebo (Arm 1)
Combination Product: CD388 — CD388 liquid for injection
  Arms: CD388 High Dose (Arm 2); CD388 Low Dose 1 (Arm 3); CD388 Low Dose 2 (Optional Arm 4); CD388 Low Dose 3 (Optional Arm 5); CD388 Low Dose 4 (Optional Arm 6)

SUMMARY:
The purpose of this study is to evaluate the preventative antiviral activity of CD388, as compared to saline placebo, when administered as a single dose to healthy adult participants in a human viral challenge model of influenza.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, proof-of-concept study in healthy adult male and female participants 18 to 55 years of age, inclusive. The primary goal of this Phase 2a study is to assess the prophylactic antiviral activity against influenza, safety, tolerability, and pharmacokinetics (PK) of CD388 via a human viral challenge (HVC) model, and to explore the impact of dose levels on efficacy. Each participant will receive a single administration of CD388 or placebo; multiple dose levels of CD388 may be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated by the participant and the PI/investigator obtained before any assessment is performed.
2. Adult male or female aged between 18 and 55 years old, inclusive, on the day prior to signing the consent form.
3. A total body weight ≥50 kilograms (kg) and body mass index (BMI) ≥18 kg/meter squared (m^2) and ≤35kg/m^2.
4. In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety, as defined by medical history, physical examination (including vital signs), electrocardiogram (ECG), and routine laboratory tests as determined by the Principal Investigator (PI)/investigator.
5. Participants will have a documented medical history either prior to entering the study or following medical history review with the study physician at screening.
6. The following criteria are applicable to female participants participating in the study.

   1. Females of childbearing potential must have a negative pregnancy test prior to enrolment.
   2. Females of non-childbearing potential:

      1. Postmenopausal females defined as amenorrhea for ≥12 months with no alternative medical cause. A high follicle-stimulating hormone (FSH) level, within appropriate postmenopausal range, may be used to confirm postmenopausal state in the absence of combined hormonal contraception or hormone replacement therapy. If there is <12 months of amenorrhea 2 FSH samples are required at least 4 to 6 weeks apart.
      2. Documented status as being surgically sterile (e.g., tubal ligation, hysterectomy, bilateral salpingectomy, and bilateral oophorectomy).
7. The following criteria apply to female and male participants:

   1. Female participants of childbearing potential must use 1 form of highly effective contraception. Hormonal methods must be in place from at least 2 weeks prior to the first study visit. The contraception use must continue until 5 effective half-lives (205 days) after the last dose of investigational medicinal product (IMP). Highly effective contraception is as described below:

      1. Established use of hormonal methods of contraception described below (for a minimum of 30 days prior to the first study visit). When hormonal methods of contraception are used, male partners are required to use a condom with a spermicide:

         * a) combined (estrogen- and progestogen containing) hormonal contraception associated with inhibition of ovulation:

           * (i) oral
           * (ii) intravaginal
           * (iii) transdermal
         * b) progestogen-only hormonal contraception associated with inhibition of ovulation:

           * (i) oral
           * (ii) injectable
           * (iii) implantable
      2. Intrauterine device.
      3. Intrauterine hormone-releasing system.
      4. Bilateral tubal ligation.
      5. Male sterilization (with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate) where the vasectomized male is the sole partner for that woman.
      6. True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant.
   2. Male participants must agree to the contraceptive requirements below at entry to quarantine and continuing until 5 effective half-lives (205 days) after the last dose of IMP.

      1. Use a condom with a spermicide to prevent pregnancy in a female partner or to prevent exposure of any partner (male or female) to the IMP.
      2. Male sterilization with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate (please note that the use of condom with spermicide will still be required to prevent partner exposure). This applies only to males participating in the study.
      3. In addition, for female partners of childbearing potential, that partner must use another form of contraception such as one of the highly effective methods mentioned above for female participants.
      4. True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant.
   3. In addition to the contraceptive requirements above, male participants must agree not to donate sperm following discharge from quarantine until 5 effective half-lives (205 days) after the last dose of IMP.
8. Sero-suitable for the challenge virus. A participant must be sero-suitable to take part in the study, i.e., he/she must have no or low pre-existing serum levels of antibodies specific to the challenge agent. Serology testing will be carried out by a hemagglutination inhibitory assay to determine serum antibody titers. As an example, a participant is considered sero-suitable if their serology (hemagglutination inhibition [HAI]) titer result is ≤10.

Exclusion Criteria:

1. History of, or currently active, symptoms or signs suggestive of upper respiratory tract (URT) or lower respiratory tract (LRT) infection within 4 weeks prior to the first study visit.
2. Any history or evidence of any clinically significant or currently active cardiovascular, respiratory, dermatological, gastrointestinal, endocrinological, hematological, hepatic, immunological (including immunosuppression), metabolic, urological, renal, neurological, or psychiatric disease and/or other major disease that, in the opinion of the PI/investigator may interfere with a participant completing the study and necessary investigations. The following conditions apply:

   1. Participants with a history of resolved depression and/or anxiety 1 or more years ago can be included if the Patient Health Questionnaire (PHQ-9) and the Generalized Anxiety Disorder Questionnaire (GAD-7) is less than or equal to 4 on admission. Participants with a history of stress-related illness, which is not ongoing or requiring current therapy, with good evidence of preceding stressors may be included at the PI's discretion. As required, participants will be assessed prior to enrolment with a PHQ-9 and GAD-7 questionnaire.
   2. Rhinitis (including hay fever) which is clinically active or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days of admission to quarantine will be excluded. Participants with a history of currently inactive rhinitis (within the last 30 days) or mild rhinitis may be included at the PI's discretion.
   3. Atopic dermatitis/eczema which is clinically severe and/or requiring moderate to large amounts of daily dermal corticosteroids will be excluded. Participants with mild to moderate atopic dermatitis/eczema, taking small amounts of regular dermal corticosteroids may be included at the PI's discretion.
   4. Any concurrent serious illness, including history of malignancy, that may interfere with a participant completing the study. Basal cell carcinoma within 5 years of initial diagnosis or with evidence of recurrence is also an exclusion.
   5. Participants reporting physician-diagnosed migraine can be included provided there are no associated neurological symptoms such as hemiplegia or visual loss. Cluster headache/migraine or prophylactic treatment for migraine is an exclusion.
   6. Participants with physician diagnosed mild irritable bowel syndrome not requiring regular treatment can be included at the discretion of the PI.
   7. Participants with a history of asthma where their last symptoms/treatment were in adolescence and over 6 years ago may be included at the discretion of the PI. Any participants with symptoms or treatment in adulthood would be excluded.
3. Any participants who have smoked ≥10 pack years at any time (10 pack years is equivalent to 1 pack of 20 cigarettes a day for 10 years).
4. Females who:

   1. Are breastfeeding, or
   2. Have been pregnant within 6 months prior to the study, or
   3. Have a positive pregnancy test at any point during screening or prior to dosing with IMP.
5. Lifetime history of anaphylaxis and/or a history of severe allergic reaction or significant intolerance to any food or drug in the last 12 months, as assessed by the PI.
6. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
7. . .

   1. Any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the aims of the study and, in particular, any of the nasal assessments or viral challenge (historical nasal polyps can be included, but large nasal polyps causing current and significant symptoms and/or requiring regular treatments in the last month will be excluded).
   2. Any clinically significant history of epistaxis (large nosebleeds) within the last 3 months of the first study visit and/or history of being hospitalized due to epistaxis on any previous occasion.
   3. Any nasal or sinus surgery within 3 months of the first study visit.
8. . .

   1. Evidence of vaccinations within the 4 weeks prior to the planned date of dosing with IMP.
   2. Intention to receive any vaccination(s) before the last day of follow-up (with the exception of vaccinations recommended for Coronavirus Disease 2019 [COVID-19] as defined by Medicines and Healthcare products Regulatory Agency (MHRA)/government vaccination guidelines).
   3. No travel restrictions apply after the Day 28 [±3 days] follow-up visit; however, we expect participants to be available to attend the clinic at the Day 60, Day 120, and Day 180 follow-up visits.
   4. Receipt of influenza vaccine in the last 6 months prior to the planned date of viral challenge.
9. Receipt of blood or blood products, or loss (including blood donations) of 550 milliliters (mL) or more of blood during the 3 months prior to the planned dosing with IMP or planned during the 3 months after the final visit.
10. . .

    1. Receipt of any investigational drug within 3 months prior to the planned date of dosing with IMP.
    2. Receipt of 3 or more investigational drugs within the previous 12 months prior to the planned date of dosing with IMP.
    3. Prior inoculation with a virus from the same virus-family as the challenge virus.
    4. Prior participation in another human viral challenge (HVC) study with a respiratory virus in the preceding 3 months, taken from the date of viral challenge in the previous study to the date of expected viral challenge in this study.
11. Use or anticipated use during the conduct of the study of concomitant medications (prescription and/or non-prescription), including vitamins or herbal and dietary supplements within the specified windows, unless in the opinion of the study physician/PI, the medication will not interfere with the study procedures or compromise participant safety. Specifically, the following are excluded:

    1. Herbal supplements within 7 days prior to the planned date of dosing with IMP.
    2. Chronically used medications, vitamins, or dietary supplements within 21 days prior to the planned date of dosing with IMP.
    3. Over-the-counter medications (e.g., paracetamol or ibuprofen) where the dose taken over the preceding 7 days prior to the planned date dosing with IMP has exceeded the maximum permissible 24-hour dose (e.g., ≥4 grams paracetamol over the preceding week).
    4. Systemic antiviral administration within 4 weeks of the planned date of dosing with IMP.
12. . .

    1. Confirmed positive test for drugs of misuse and cotinine on first study visit. One repeat test is allowed at PI discretion.
    2. Recent history or presence of alcohol addiction, or excessive use of alcohol (weekly intake in excess of 28 units alcohol; 1 unit being a half glass of beer, a small glass of wine, or a measure of spirits), or excessive consumption of xanthine-containing substances (e.g., daily intake in excess of 5 cups of caffeinated drinks, e.g., coffee, tea, cola).
13. A forced expiratory volume in 1 second (FEV1) <80 percent.
14. Positive human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) test (HIV positive - via 3 confirmatory tests - Vidas, Genenius, and Determine; HBV confirmed via hepatitis B surface antigen [HbsAG], hepatitis B surface antibody [anti-HBs], and hepatitis B core antibody [anti-HBc] [immunoglobulin G/immunoglobulin M]; and HCV confirmed via hepatitis C viral load).
15. Presence of fever, defined as participant presenting with a temperature reading of ≥37.9 degrees Celsius (°C) on Day -7/-6 and/or pre-dose on Day -5.
16. Those employed or immediate relatives of those employed at hVIVO Services Limited (hVIVO) or the sponsor.
17. Any other finding that, in the opinion of the PI/investigator, deems the participant unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Equils, MD, Study Director — Cidara Therapeutics Inc.; Arun Anandakumar, MD, Principal Investigator — hVIVO Services Limited
Locations (1):
- hVIVO Services Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rojas RE, Equils O, Villacian J, Mann A, van Duijnhoven W, Vingerhoets J, Baguet T, Wang SS, Anandakumar A, Anger A, Tourneroche A, Silva IG, Flanagan S. Prophylactic Efficacy of CD388, a Novel Drug-Fc Conjugate, in a Human Influenza A/H3N2 Virus Challenge Model: A Randomized, Controlled Phase 2a Study. Clin Infect Dis. 2025 Dec 24;81(5):e310-e318. doi: 10.1093/cid/ciaf465. PMID 41060047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 168 participants in up to 2 cohorts were planned for enrollment in the study. Due to low participant eligibility, the randomization schedule was changed in Cohort 1 after the first quarantine group to only randomize participants to the 150 mg CD388 and placebo arms. With only 2 participants in the 50 mg CD388 arm, safety and demographic data only have been reported. Based on data from the planned interim analysis of Cohort 1, a decision was made to not proceed with Cohort 2.
Groups:
- Placebo: Up to 30 participants randomized to receive a single dose of saline placebo, administered by subcutaneous (SQ) injection, prior to being inoculated with the influenza challenge virus
  Saline placebo: Sterile normal saline for injection
- 50 mg CD388: Up to 30 participants randomized to receive a single dose of 50 milligrams (mg) CD388, administered by SQ injection, prior to being inoculated with the influenza challenge virus
  CD388: CD388 liquid for injection
- 150 mg CD388: Up to 30 participants randomized to receive a single dose of 150 mg CD388, administered by SQ injection, prior to being inoculated with the influenza challenge virus
  CD388: CD388 liquid for injection
Period: Overall Study
Arm/Group | Placebo | 50 mg CD388 | 150 mg CD388
Started (All participants received their assigned treatment, and all but 1 participant in the placebo arm received challenge virus.) | 29 | 2 | 28
Completed (Two participants, both in the placebo arm, discontinued the study prior to completion. For all other participants (n=57), including the participant in the placebo arm who was not inoculated with the challenge virus, the study status was reported as completed.) | 27 | 2 | 28
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg CD388 | 150 mg CD388 | Total
Number analyzed (Participants) | 29 | 2 | 28 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.03 (8.21) | 27.50 (2.12) | 33.82 (7.86) | 33.22 (7.92)
Age, Continuous [Median (Full Range); unit: years] | 31.00 [22.0 to 51.0] | 27.50 [26.0 to 29.0] | 32.00 [21.0 to 51.0] | 31.00 [21.0 to 51.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 13 | 22
  Male | 20 | 2 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 2 | 28 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4
  White | 24 | 1 | 23 | 48
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 29 | 2 | 28 | 59
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 76.29 (13.26) | 72.40 (2.55) | 79.68 (19.02) | 77.77 (16.04)
Weight [Median (Full Range); unit: kg] | 72.90 [54.2 to 100.8] | 72.40 [70.6 to 74.2] | 75.60 [54.2 to 112.0] | 75.20 [54.2 to 112.0]
Height [Mean (Standard Deviation); unit: meters (m)] | 1.72 (0.08) | 1.70 (0.11) | 1.74 (0.09) | 1.73 (0.09)
Height [Median (Full Range); unit: meters (m)] | 1.72 [1.6 to 1.9] | 1.70 [1.6 to 1.8] | 1.77 [1.6 to 1.9] | 1.74 [1.6 to 1.9]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meter^2 (kg/m^2)] | 25.63 (3.49) | 25.15 (2.47) | 26.09 (4.45) | 25.83 (3.91)
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 25.00 [21.1 to 31.4] | 25.15 [23.4 to 26.9] | 24.60 [20.5 to 33.8] | 24.90 [20.5 to 33.8]

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Viral Load-Time Curve (VL-AUC) After Influenza Viral Challenge
Description: Evaluation of the prophylactic effect of CD388, when compared to placebo, on VL-AUC of influenza challenge virus as determined by quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR) on nasal samples starting 1 day post viral challenge.
Time Frame: Day 1 (evening [pm]); Days 2, 3, 4, 5, 6, and 7 (morning [am] and pm); Day 8 (am)
Population: The Per-Protocol Population included all randomized participants who received at least 1 dose of study intervention and were challenged with the study virus, and who have a valid result for at least 80% of the planned qRT-PCR nasal samples from Day 1 (pm) up to Day 8 (am) (i.e., at least 11 out of 14), and who present no major deviations likely to impact the evaluation of the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: log[10] copies/milliliter (mL)*hour
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
log[10] copies/milliliter (mL)*hour | 16.09 (11.86) | 10.70 (8.01)
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.0390, Wilcoxon (Mann-Whitney) — alpha = 0.025 one-sided; Hodges-Lehmann estimator = -1.2, 95% CI 2-sided [-5.7 to 0.0]

2. Primary Outcome: Median Area Under the Viral Load-Time Curve (VL-AUC) After Influenza Viral Challenge
Description: as for outcome 1
Time Frame: Day 1 (evening [pm]); Days 2, 3, 4, 5, 6, and 7 (morning [am] and pm); Day 8 (am)
Population: as for outcome 1
Measure: Median (Full Range); unit: log[10] copies/mL*hour
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
log[10] copies/mL*hour | 8.52 [6.4 to 39.8] | 6.40 [6.4 to 29.9]

3. Secondary Outcome: Mean Peak Viral Load by qRT-PCR After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the peak (i.e., maximum) viral load of influenza as determined by quantifiable qRT-PCR measurements in nasal samples starting 1 day post viral challenge.
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log[10] copies/mL
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
log[10] copies/mL | 4.28 (2.94) | 2.84 (2.40)
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.0185, Wilcoxon (Mann-Whitney) — alpha = 0.025 one-sided; Mean Difference (Net) = -1.4, 95% CI 2-sided [-2.9 to -0.0]

4. Secondary Outcome: Median Peak Viral Load by qRT-PCR After Influenza Viral Challenge
Description: as for outcome 3
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Median (Full Range); unit: log[10] copies/mL
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
log[10] copies/mL | 3.79 [1.0 to 8.5] | 0.97 [0.9 to 7.5]

5. Secondary Outcome: Time to Confirmed Negative Test by qRT-PCR After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the time (in hours, as estimated using the Kaplan-Meier method) to confirmed negative test for influenza as determined by quantifiable qRT-PCR measurements in nasal samples starting 1 day post viral challenge.
Time Frame: From Day 1 (pm) until the first confirmed undetectable assessment after peak measurement, assessed up to Day 8 (am)
Population: The Per-Protocol Population included all randomized participants who received at least 1 dose of study intervention and were challenged with the study virus, and who have a valid result for at least 80% of the planned qRT-PCR nasal samples from Day 1 (pm) up to Day 8 (am) (i.e., at least 11 out of 14), and who present no major deviations likely to impact the evaluation of the primary efficacy endpoint. NOTE: Participants without a detectable qRT-PCR value were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: hours
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 19 | 12
hours
  25th Percentile | 61.9 [14.7 to 120.3] | 66.7 [24.3 to 72.4]
  Median | 134.1 [61.9 to NA] — Some values were not computable due to the lack of an event {i.e., the first result equal to not detected (less than the Lower Level of Detection [<LLOD]) after peak measure} at the assessed timepoint. | 79.4 [24.4 to 143.1]
  75th Percentile | 158.3 [134.1 to NA] — Some values were not computable due to the lack of an event {i.e., the first result equal to not detected (less than the Lower Level of Detection [<LLOD]) after peak measure} at the assessed timepoint. | 131.7 [72.4 to NA] — Some values were not computable due to the lack of an event {i.e., the first result equal to not detected (less than the Lower Level of Detection [<LLOD]) after peak measure} at the assessed timepoint.
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.0613, Gehan-Wilcoxon — alpha = 0.025 one-sided

6. Secondary Outcome: Mean Area Under the Viral Load-Time Curve (VL-AUC) by Viral Culture After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on VL-AUC of influenza challenge virus as determined by viral culture on nasal samples starting 1 day post viral challenge.
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log[10] copies/mL*hour
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
log[10] copies/mL*hour | 5.82 (3.70) | 3.95 (1.57)
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.1587, Wilcoxon (Mann-Whitney) — alpha = 0.025 one-sided; Hodges-Lehmann estimator = -0.0, 95% CI 2-sided [-2.4 to 0.0]

7. Secondary Outcome: Median Area Under the Viral Load-Time Curve (VL-AUC) by Viral Culture After Influenza Viral Challenge
Description: as for outcome 6
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Median (Full Range); unit: log[10] copies/mL*hour
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
log[10] copies/mL*hour | 3.29 [3.2 to 14.4] | 3.29 [3.2 to 9.7]

8. Secondary Outcome: Mean Peak Viral Load by Viral Culture After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the peak (i.e., maximum) viral load of influenza as determined by quantitative viral culture measurements in nasal samples starting 1 day post viral challenge.
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log[10] copies/mL
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
log[10] copies/mL | 2.13 (2.10) | 1.07 (1.18)
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.0236, Wilcoxon (Mann-Whitney) — alpha = 0.025 one-sided; Mean Difference (Net) = -1.1, 95% CI 2-sided [-2.0 to -0.1]

9. Secondary Outcome: Median Peak Viral Load by Viral Culture After Influenza Viral Challenge
Description: as for outcome 8
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Median (Full Range); unit: log[10] copies/mL
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
log[10] copies/mL | 0.50 [0.5 to 5.5] | 0.50 [0.5 to 4.5]

10. Secondary Outcome: Time to Confirmed Negative Test by Viral Culture After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the time (in hours, as estimated using the Kaplan-Meier method) to confirmed negative test for influenza as determined by quantifiable viral culture measurements in nasal samples starting 1 day post viral challenge.
Time Frame: From Day 1 (pm) until the first confirmed undetectable assessment after peak measurement, assessed up to Day 8 (am)
Population: The Per-Protocol Population included all randomized participants who received at least 1 dose of study intervention and were challenged with the study virus, and who have a valid result for at least 80% of the planned qRT-PCR nasal samples from Day 1 (pm) up to Day 8 (am) (i.e., at least 11 out of 14), and who present no major deviations likely to impact the evaluation of the primary efficacy endpoint. NOTE: Participants without a detectable viral culture value were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: hours
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 11 | 6
hours
  25th Percentile | 71.4 [47.2 to 85.9] | 62.3 [24.3 to 85.9]
  Median | 85.9 [47.5 to 110.1] | 78.7 [24.3 to NA] — Some values were not computable due to the lack of an event {i.e., the first result equal to not detected (less than the Lower Level of Detection [<LLOD]) after peak measure} at the assessed timepoint.
  75th Percentile | 110.1 [85.9 to NA] — Some values were not computable due to the lack of an event {i.e., the first result equal to not detected (less than the Lower Level of Detection [<LLOD]) after peak measure} at the assessed timepoint. | 86.0 [62.3 to NA] — Some values were not computable due to the lack of an event {i.e., the first result equal to not detected (less than the Lower Level of Detection [<LLOD]) after peak measure} at the assessed timepoint.
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.1282, Gehan-Wilcoxon — alpha = 0.025 one-sided

11. Secondary Outcome: Mean Area Under the Total Clinical Symptoms Score-Time Curve (TSS-AUC) After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on TSS-AUC as measured by graded symptom scoring system (participant completed symptom diary card) collected 3 times daily starting 1 day post viral challenge.
  At each assessment, the participant provides scores from 0 to 3 for a list of 13 symptoms (runny nose, stuffy nose, sneezing, sore throat, earache, malaise/tiredness, headache, muscle and/or joint ache, chilliness/feverishness, cough, chest tightness, shortness of breath, and wheeze). Grade 0: no symptoms; grade 1: just noticeable; grade 2: clearly bothersome from time to time but does not interfere with normal daily activities; grade 3: quite bothersome most or all the time and stops participation in activities.
  An individual Total Symptom Score (TSS) is derived at each assessment of the diary card as the sum of the scores given to the 13 symptoms on that symptom score card, resulting in possible TSS values from 0 to 39.
Time Frame: Three (3) times per day, at the same time each day (±1 hour), on Days 1, 2, 3, 4, 5, 6, and 7; and on Day 8 (am only)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: TSS points*day
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
TSS points*day | 7.66 (14.13) | 2.22 (4.86)
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.2877, Wilcoxon (Mann-Whitney) — alpha = 0.025 one-sided; Mean Difference (Net) = -5.4, 95% CI 2-sided [-11.2 to 0.3]

12. Secondary Outcome: Median Area Under the Total Clinical Symptoms Score-Time Curve (TSS-AUC) After Influenza Viral Challenge
Description: as for outcome 11
Time Frame: Three (3) times per day, at the same time each day (±1 hour), on Days 1, 2, 3, 4, 5, 6, and 7; and on Day 8 (am only)
Population: as for outcome 1
Measure: Median (Full Range); unit: TSS points*day
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
TSS points*day | 0.45 [0.0 to 48.3] | 0.86 [0.0 to 25.2]

13. Secondary Outcome: Mean Peak Total Clinical Symptoms Score (TSS) After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the peak (i.e., maximum) TSS score as measured by graded symptom scoring system (participant completed symptom diary card) collected 3 times daily starting 1 day post viral challenge.
  At each assessment, the participant provides scores from 0 to 3 for a list of 13 symptoms (runny nose, stuffy nose, sneezing, sore throat, earache, malaise/tiredness, headache, muscle and/or joint ache, chilliness/feverishness, cough, chest tightness, shortness of breath, and wheeze). Grade 0: no symptoms; grade 1: just noticeable; grade 2: clearly bothersome from time to time but does not interfere with normal daily activities; grade 3: quite bothersome most or all the time and stops participation in activities.
  An individual Total Symptom Score (TSS) is derived at each assessment of the diary card as the sum of the scores given to the 13 symptoms on that symptom score card, resulting in possible TSS values from 0 to 39.
Time Frame: Three (3) times per day, at the same time each day (±1 hour), on Days 1, 2, 3, 4, 5, 6, and 7; and on Day 8 (am only)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: total symptom score
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
total symptom score | 3.54 (5.34) | 1.79 (3.12)
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.2517, Wilcoxon (Mann-Whitney) — alpha = 0.025 one-sided; Mean Difference (Net) = -1.8, 95% CI 2-sided [-4.1 to 0.6]

14. Secondary Outcome: Median Peak Total Clinical Symptoms Score (TSS) After Influenza Viral Challenge
Description: as for outcome 13
Time Frame: Three (3) times per day, at the same time each day (±1 hour), on Days 1, 2, 3, 4, 5, 6, and 7; and on Day 8 (am only)
Population: as for outcome 1
Measure: Median (Full Range); unit: total symptom score
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
total symptom score | 1.00 [0.0 to 21.0] | 1.00 [0.0 to 16.0]

15. Secondary Outcome: Mean Individual Peak Daily Total Clinical Symptoms Score After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the peak (i.e., maximum) daily symptom score (i.e., individual maximum daily sum of symptom score) as measured by graded symptom scoring system (participant completed symptom diary card) collected 3 times daily starting 1 day post viral challenge.
  At each assessment, the participant provides scores from 0 to 3 for a list of 13 symptoms (runny nose, stuffy nose, sneezing, sore throat, earache, malaise/tiredness, headache, muscle and/or joint ache, chilliness/feverishness, cough, chest tightness, shortness of breath, and wheeze). Grade 0: no symptoms; grade 1: just noticeable; grade 2: clearly bothersome from time to time but does not interfere with normal daily activities; grade 3: quite bothersome most or all the time and stops participation in activities.
  An individual Total Symptom Score (TSS) is derived at each assessment as the sum of the scores given to the 13 symptoms, giving possible TSS values from 0 to 39.
Time Frame: From Day 1 up to Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: total symptom score
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
total symptom score
  Quarantine Day 1 | 0.64 (1.50) | 0.46 (0.84)
  Quarantine Day 2 | 2.29 (4.60) | 0.75 (2.12)
  Quarantine Day 3 | 2.79 (5.10) | 1.25 (3.15)
  Quarantine Day 4 | 2.11 (3.83) | 0.82 (1.85)
  Quarantine Day 5 | 1.07 (2.12) | 0.36 (0.87)
  Quarantine Day 6 | 0.79 (1.91) | 0.39 (0.69)
  Quarantine Day 7 | 0.43 (1.53) | 0.07 (0.26)
  Quarantine Day 8 Discharge | 0.15 (0.60) | 0.11 (0.42)

16. Secondary Outcome: Median Individual Peak Daily Total Clinical Symptoms Score After Influenza Viral Challenge
Description: as for outcome 15
Time Frame: From Day 1 up to Day 8
Population: as for outcome 1
Measure: Median (Full Range); unit: total symptom score
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
total symptom score
  Quarantine Day 1 | 0.00 [0.0 to 7.0] | 0.00 [0.0 to 3.0]
  Quarantine Day 2 | 0.00 [0.0 to 17.0] | 0.00 [0.0 to 11.0]
  Quarantine Day 3 | 0.00 [0.0 to 21.0] | 0.00 [0.0 to 16.0]
  Quarantine Day 4 | 0.00 [0.0 to 14.0] | 0.00 [0.0 to 8.0]
  Quarantine Day 5 | 0.00 [0.0 to 8.0] | 0.00 [0.0 to 4.0]
  Quarantine Day 6 | 0.00 [0.0 to 9.0] | 0.00 [0.0 to 2.0]
  Quarantine Day 7 | 0.00 [0.0 to 8.0] | 0.00 [0.0 to 1.0]
  Quarantine Day 8 Discharge | 0.00 [0.0 to 3.0] | 0.00 [0.0 to 2.0]

17. Secondary Outcome: Time to Symptom Resolution After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the time (in hours, as estimated using the Kaplan-Meier method) to symptom resolution (i.e., first time with Total Symptom Score [TSS] equal to the TSS at baseline after which no further increase above the baseline TSS was observed) as measured by graded daily symptom scoring system (participant completed symptom diary card) collected 3 times daily starting 1 day post viral challenge.
  An individual TSS is derived at each assessment of the diary card as the sum of the scores given to the 13 symptoms on that symptom score card, resulting in possible TSS values from 0 to 39.
Time Frame: Starting Day 1, from the time of peak daily symptom score until the time of returning to baseline score, up to Day 8
Population: The Per-Protocol Population included all randomized participants who received at least 1 dose of study intervention and were challenged with the study virus, and who have a valid result for at least 80% of the planned qRT-PCR nasal samples from Day 1 (pm) up to Day 8 (am) (i.e., at least 11 out of 14), and who present no major deviations likely to impact the evaluation of the primary efficacy endpoint. NOTE: Participants who only had a baseline TSS were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: hours
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 19 | 18
hours
  25th Percentile | 8.4 [6.9 to 31.1] | 23.3 [6.7 to 54.3]
  Median | 41.5 [8.4 to 72.7] | 74.8 [23.3 to 96.2]
  75th Percentile | 78.7 [41.5 to NA] — Some values were not computable due to the lack of an event at the assessed timepoint. | 133.5 [84.4 to NA] — Some values were not computable due to the lack of an event at the assessed timepoint.
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.9024, Gehan-Wilcoxon — alpha = 0.025 one-sided

18. Secondary Outcome: Number of Participants With qRT-PCR-Confirmed Influenza Infection After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the number of participants with qRT-PCR-confirmed influenza infection, defined as 2 quantifiable (≥ lower limit of quantification [LLOQ]) qRT-PCR measurements (reported on 2 or more independent nasal samples over 2 days), starting 1 day post viral challenge.
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
Participants
  No qRT-PCR-confirmed Influenza Infection | 14 | 22
  qRT-PCR-confirmed Influenza Infection | 14 | 6
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.0248, Fisher Exact — alpha = 0.025 one-sided

19. Secondary Outcome: Percentage of Participants With qRT-PCR-Confirmed Influenza Infection After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the percentage of participants with qRT-PCR-confirmed influenza infection, defined as 2 quantifiable (≥ lower limit of quantification [LLOQ]) qRT-PCR measurements (reported on 2 or more independent nasal samples over 2 days), starting 1 day post viral challenge.
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
percentage of participants
  No qRT-PCR-confirmed Influenza Infection | 50.0 [30.6 to 69.4] | 78.6 [59.0 to 91.7]
  qRT-PCR-confirmed Influenza Infection | 50.0 [30.6 to 69.4] | 21.4 [8.3 to 41.0]

20. Secondary Outcome: Number of Participants With at Least One Positive Quantitative (≥LLOQ) Cell Culture After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the number of participants with at least 1 positive quantitative (≥LLOQ) cell culture measurement in nasal samples starting 1 day post viral challenge.
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
Participants
  No Positive Quantitative (≥LLOQ) Cell Culture | 17 | 22
  At Least 1 Positive Quantitative (≥LLOQ) Cell Culture | 11 | 6
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.1224, Fisher Exact — alpha = 0.025 one-sided

21. Secondary Outcome: Percentage of Participants With at Least One Positive Quantitative (≥LLOQ) Cell Culture After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the percentage of participants with at least 1 positive quantitative (≥LLOQ) cell culture measurement in nasal samples starting 1 day post viral challenge.
Time Frame: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
percentage of participants
  No Positive Quantitative (≥LLOQ) Cell Culture | 60.7 [40.6 to 78.5] | 78.6 [59.0 to 91.7]
  At Least 1 Positive Quantitative (≥LLOQ) Cell Culture | 39.3 [21.5 to 59.4] | 21.4 [8.3 to 41.0]

22. Secondary Outcome: Number of Participants With qRT-PCR-Confirmed Symptomatic Influenza Infection After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the number of participants with qRT-PCR-confirmed symptomatic influenza infection starting 1 day post viral challenge, defined as:
  * RT-PCR-confirmed influenza infection (2 quantifiable [≥LLOQ] qRT-PCR measurements [reported on 2 or more independent nasal samples over 2 days]), AND
  * TSS score ≥2 at any single time point (i.e., any individual symptom diary card for which the sum of symptom scores is ≥2; e.g., at a minimum, ≥1 symptom of grade ≥2, or ≥2 symptoms of grade ≥1), as measured by graded symptom scoring system (participant completed symptom diary card) collected 3 times daily.
Time Frame: • For qRT-PCR measurements: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am) • For TSS measurements: Three (3) times per day, at the same time each day (±1 hour), on Days 1, 2, 3, 4, 5, 6, and 7; and on Day 8 (am only)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
Participants
  No qRT-PCR-confirmed Symptomatic Influenza Infection | 19 | 24
  qRT-PCR-confirmed Symptomatic Influenza Infection | 9 | 4
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.1023, Fisher Exact — alpha = 0.025 one-sided

23. Secondary Outcome: Percentage of Participants With qRT-PCR-Confirmed Symptomatic Influenza Infection After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the percentage of participants with qRT-PCR-confirmed symptomatic influenza infection starting 1 day post viral challenge, defined as:
  * RT-PCR-confirmed influenza infection (2 quantifiable [≥LLOQ] qRT-PCR measurements [reported on 2 or more independent nasal samples over 2 days]), AND
  * TSS score ≥2 at any single time point (i.e., any individual symptom diary card for which the sum of symptom scores is ≥2; e.g., at a minimum, ≥1 symptom of grade ≥2, or ≥2 symptoms of grade ≥1), as measured by graded symptom scoring system (participant completed symptom diary card) collected 3 times daily.
Time Frame: as for outcome 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
percentage of participants
  No qRT-PCR-confirmed Symptomatic Influenza Infection | 67.9 [47.6 to 84.1] | 85.7 [67.3 to 96.0]
  qRT-PCR-confirmed Symptomatic Influenza Infection | 32.1 [15.9 to 52.4] | 14.3 [4.0 to 32.7]

24. Secondary Outcome: Number of Participants With qRT-PCR-Confirmed Moderately Severe Symptomatic Influenza Infection After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the number of participants with qRT-PCR-confirmed moderately severe symptomatic influenza infection starting 1 day post viral challenge, defined as:
  * RT-PCR-confirmed influenza infection (2 quantifiable [≥LLOQ] qRT-PCR measurements [reported on 2 or more independent nasal samples over 2 days]), AND
  * One or more symptoms of grade ≥2 at a single time point (i.e., on any individual symptom card), as measured by graded symptom scoring system (participant completed symptom diary card) collected 3 times daily.
Time Frame: • For qRT-PCR measurements: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am) • For symptom scoring measurements: Three (3) times per day, at the same time each day (±1 hour), on Days 1, 2, 3, 4, 5, 6, and 7; and on Day 8 (am only)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
Participants
  No qRT-PCR-confirmed Moderately Severe Symptomatic Influenza Infection | 21 | 25
  qRT-PCR-confirmed Moderately Severe Symptomatic Influenza Infection | 7 | 3
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.1477, Fisher Exact — alpha = 0.025 one-sided

25. Secondary Outcome: Percentage of Participants With qRT-PCR-Confirmed Moderately Severe Symptomatic Influenza Infection After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the percentage of participants with qRT-PCR-confirmed moderately severe symptomatic influenza infection starting 1 day post viral challenge, defined as:
  * RT-PCR-confirmed influenza infection (2 quantifiable [≥LLOQ] qRT-PCR measurements [reported on 2 or more independent nasal samples over 2 days]), AND
  * One or more symptoms of grade ≥2 at a single time point (i.e., on any individual symptom card), as measured by graded symptom scoring system (participant completed symptom diary card) collected 3 times daily.
Time Frame: as for outcome 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
percentage of participants
  No qRT-PCR-confirmed Moderately Severe Symptomatic Influenza Infection | 75.0 [55.1 to 89.3] | 89.3 [71.8 to 97.7]
  qRT-PCR-confirmed Moderately Severe Symptomatic Influenza Infection | 25.0 [10.7 to 44.9] | 10.7 [2.3 to 28.2]

26. Secondary Outcome: Number of Participants With Culture Lab-Confirmed Symptomatic Influenza Infection After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the number of participants with culture laboratory-confirmed symptomatic influenza infection starting 1 day post viral challenge, defined as:
  * Lab-confirmed culturable influenza infection (1 quantifiable [≥LLOQ] cell culture measurement in nasal samples), AND
  * TSS score ≥2 at any single time point (i.e., any individual symptom diary card for which the sum of symptom scores is ≥2; e.g., at a minimum, ≥1 symptom of grade ≥2, or ≥2 symptoms of grade ≥1), as measured by graded symptom scoring system (participant completed symptom diary card) collected 3 times daily.
Time Frame: • For viral culture measurements: Day 1 (pm); Days 2, 3, 4, 5, 6, and 7 (am and pm); Day 8 (am) • For TSS measurements: Three (3) times per day, at the same time each day (±1 hour), on Days 1, 2, 3, 4, 5, 6, and 7; and on Day 8 (am only)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
Participants
  No Culture Lab-confirmed Symptomatic Influenza Infection | 20 | 24
  Culture Lab-confirmed Symptomatic Influenza Infection | 8 | 4
Statistical Analysis 1: Comparison: Placebo vs 150 mg CD388; Test type: Superiority; p = 0.1645, Fisher Exact — alpha = 0.025 one-sided

27. Secondary Outcome: Percentage of Participants With Culture Lab-Confirmed Symptomatic Influenza Infection After Influenza Viral Challenge
Description: Evaluation of the effect of CD388, when compared to placebo, on the percentage of participants with culture laboratory-confirmed symptomatic influenza infection starting 1 day post viral challenge, defined as:
  * Lab-confirmed culturable influenza infection (1 quantifiable [≥LLOQ] cell culture measurement in nasal samples), AND
  * TSS score ≥2 at any single time point (i.e., any individual symptom diary card for which the sum of symptom scores is ≥2; e.g., at a minimum, ≥1 symptom of grade ≥2, or ≥2 symptoms of grade ≥1), as measured by graded symptom scoring system (participant completed symptom diary card) collected 3 times daily.
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 150 mg CD388
Number analyzed (Participants) | 28 | 28
percentage of participants
  No Culture Lab-confirmed Symptomatic Influenza Infection | 71.4 [51.3 to 86.8] | 85.7 [67.3 to 96.0]
  Culture Lab-confirmed Symptomatic Influenza Infection | 28.6 [13.2 to 48.7] | 14.3 [4.0 to 32.7]

28. Secondary Outcome: Occurrence of Solicited Adverse Events (AEs) From Subcutaneous (SQ) Dosing up to Viral Challenge - Number of Participants
Description: Evaluation of the occurrence of solicited AEs in participants dosed with CD388, when compared with placebo, from the time of SQ dosing up to the time of inoculation with the influenza challenge virus, based on the number of participants reporting any solicited AE.
  Solicited AEs are those predefined events relating to reactogenicity (pain, tenderness, erythema/redness, induration/swelling) for which participants were specifically questioned and which were noted by participants in a participant diary.
Time Frame: From Day -5 (dosing) up to Day 0 (viral challenge)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg CD388 | 150 mg CD388
Number analyzed (Participants) | 28 | 2 | 28
Participants | 0 | 0 | 1

29. Secondary Outcome: Occurrence of Solicited Adverse Events (AEs) From Subcutaneous (SQ) Dosing up to Viral Challenge - Number of Events
Description: Evaluation of the occurrence of solicited AEs in participants dosed with CD388, when compared with placebo, from the time of SQ dosing up to the time of inoculation with the influenza challenge virus, based on the number of events reported.
  Solicited AEs are those predefined events relating to reactogenicity (pain, tenderness, erythema/redness, induration/swelling) for which participants were specifically questioned and which were noted by participants in a participant diary.
Time Frame: From Day -5 (dosing) up to Day 0 (viral challenge)
Population: as for baseline characteristics
Measure: Number; unit: events
Arm/Group | Placebo | 50 mg CD388 | 150 mg CD388
Number analyzed (Participants) | 28 | 2 | 28
events | 0 | 0 | 1

30. Secondary Outcome: Occurrence of Unsolicited AEs From SQ Dosing up to Day 28 Follow-up Visit - Number of Participants
Description: Evaluation of the occurrence of unsolicited AEs in participants dosed with CD388, when compared with placebo, from the time of SQ dosing up to the time of the Day 28 follow-up visit, based on the number of participants for whom any AE is observed.
  Unsolicited AEs are any AEs observed by the participant or Principal Investigator (PI)/investigator which are not prelisted on a symptom diary card.
  Results are categorized by period:
  * Period 1 (from Day -5 dosing to just before challenge virus inoculation on Day 0)
  * Period 2 (from Day 0 challenge virus inoculation to actual discharge from the quarantine unit [as scheduled on Day 8 or later at PI's decision])
  * Period 3 (from actual discharge from the quarantine unit to Day 28 (±3 days)
Time Frame: From Day -5 (dosing) up to Day 28 (±3 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg CD388 | 150 mg CD388
Number analyzed (Participants) | 29 | 2 | 28
Participants
  Period 1 | 1 | 1 | 0
  Periods 1 and 2 | 4 | 1 | 2
  Period 2 | 3 | 1 | 2
  Periods 2 and 3 | 10 | 1 | 11
  Period 3 | 8 | 1 | 9

31. Secondary Outcome: Occurrence of Unsolicited AEs From SQ Dosing up to Day 28 Follow-up Visit - Number of Events
Description: Evaluation of the occurrence of unsolicited AEs in participants dosed with CD388, when compared with placebo, from the time of SQ dosing up to the time of the Day 28 follow-up visit, based on the number of events reported.
  Unsolicited AEs are any AEs observed by the participant or Principal Investigator (PI)/investigator which are not prelisted on a symptom diary card.
  Results are categorized by period:
  * Period 1 (from Day -5 dosing to just before challenge virus inoculation on Day 0)
  * Period 2 (from Day 0 challenge virus inoculation to actual discharge from the quarantine unit [as scheduled on Day 8 or later at PI's decision])
  * Period 3 (from actual discharge from the quarantine unit to Day 28 (±3 days)
Time Frame: From Day -5 (dosing) up to Day 28 (±3 days)
Population: as for baseline characteristics
Measure: Number; unit: events
Arm/Group | Placebo | 50 mg CD388 | 150 mg CD388
Number analyzed (Participants) | 29 | 2 | 28
events
  Period 1 | 1 | 1 | 0
  Periods 1 and 2 | 4 | 2 | 2
  Period 2 | 3 | 1 | 2
  Periods 2 and 3 | 12 | 3 | 13
  Period 3 | 9 | 2 | 11

32. Secondary Outcome: Occurrence of Unsolicited AEs From SQ Dosing up to the Final Follow-up Visit - Number of Participants
Description: Evaluation of the occurrence of unsolicited AEs in participants dosed with CD388, when compared with placebo, from the time of SQ dosing up to the time of the Day 180 final follow-up visit, based on the number of participants for whom any AE was observed.
  Unsolicited AEs are any AEs observed by the participant or Principal Investigator (PI)/investigator which are not prelisted on a symptom diary card.
  Results are categorized by period:
  * Period 3 (from actual discharge from the quarantine unit to Day 28 [±3 days])
  * Period 4 (from Day 28[±3 days] to the final follow-up visit [Day 180 ±14 days])
  * Across All Periods (from Day -5 dosing to the final follow-up visit [Day 180 ±14 days])
Time Frame: From Day -5 (dosing) up to Day 180 (±14 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg CD388 | 150 mg CD388
Number analyzed (Participants) | 29 | 2 | 28
Participants
  Period 3 | 8 | 1 | 9
  Periods 3 and 4 | 16 | 1 | 19
  Period 4 | 9 | 0 | 14
  Across All Periods | 19 | 1 | 21

33. Secondary Outcome: Occurrence of Unsolicited AEs From SQ Dosing up to the Final Follow-up Visit - Number of Events
Description: Evaluation of the occurrence of unsolicited AEs in participants dosed with CD388, when compared with placebo, from the time of SQ dosing up to the time of the Day 180 final follow-up visit, based on the number of events reported.
  Unsolicited AEs are any AEs observed by the participant or Principal Investigator (PI)/investigator which are not prelisted on a symptom diary card.
  Results are categorized by period:
  * Period 3 (from actual discharge from the quarantine unit to Day 28 [±3 days])
  * Period 4 (from Day 28[±3 days] to the final follow-up visit [Day 180 ±14 days])
  * Across All Periods (from Day -5 dosing to the final follow-up visit [Day 180 ±14 days])
Time Frame: From Day -5 (dosing) up to Day 180 (±14 days)
Population: as for baseline characteristics
Measure: Number; unit: events
Arm/Group | Placebo | 50 mg CD388 | 150 mg CD388
Number analyzed (Participants) | 29 | 2 | 28
events
  Period 3 | 9 | 2 | 11
  Periods 3 and 4 | 21 | 2 | 32
  Period 4 | 12 | 0 | 21
  Across All Periods | 25 | 4 | 34

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for all participants from the time of signing the study-specific informed consent form until the last scheduled follow-up visit (Day 180 ±14 days).
Description: For evaluation purposes, two categories of AE were defined:
  * Solicited AE: predefined events relating to reactogenicity (pain, tenderness, erythema/redness, induration/swelling) for which participants were specifically questioned and which were noted by participants in a participant diary.
  * Unsolicited AE: any AEs observed by the participant or Principal Investigator (PI)/investigator which are not prelisted on a symptom diary card.
Groups:
- All Arms: The combined total of participants from all arms (Placebo, 50 mg CD388, and 150 mg CD388)
Arm/Group | Placebo | 50 mg CD388 | 150 mg CD388 | All Arms
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/2 | 0/28 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/2 | 0/28 | 0/59
Other Adverse Events (participants affected / at risk) | 19/29 | 1/2 | 21/28 | 41/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | 50 mg CD388 (N=2) | 150 mg CD388 (N=28) | All Arms (N=59)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 12 (14) | 1 (1) | 15 (19) | 28 (34)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Electrocardiogram T-wave inversion (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT05523089/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT05523089/SAP_001.pdf